CLINICAL TRIAL: NCT02269696
Title: The Effect of Metoprolol on Anaesthesia, the Need for Analgesics, and Pain in Breast Cancer Patients
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Withdrawn
Sponsor: Kuopio University Hospital (Other)
Responsible Party: Principal Investigator, Lasse Harkanen, DR, Kuopio University Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: KUH5101090
Record Dates: First submitted 2014-09-19; First posted 2014-10-21 (Estimated); Last update posted 2018-03-22 (Actual); Status verified 2018-03

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Metoprolol; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Metoprolol (Experimental): Metoprolol infusion
  Interventions: Drug: Metoprolol
- Normal saline (Placebo Comparator): Equal volume of saline.
  Interventions: Drug: Normal saline

INTERVENTIONS:
Drug: Metoprolol — Intraoperative metoprolol infusion.
  Other Names: Seloken
  Arms: Metoprolol
Drug: Normal saline — Equal of volume compared to metoprolol.
  Other Names: NaCl 0,9%
  Arms: Normal saline

SUMMARY:
The purpose of the study is to test the effects of metoprolol on anaesthesia and the need for perioperative analgesics in patients undergoing breast surgery. With 12 months follow-up the incidence of pain and life satisfaction will be evaluated.

DETAILED DESCRIPTION:
The purpose of the study is to test the effects of intraoperative metoprolol on 1) anaesthetic and alagesic use 2) pain during the early postoperative period and 3) the incidence of pain and lide satisfaction up to 12 months after the surgery. Adverse effects will be recorded as safety measures.

ELIGIBILITY:
Inclusion Criteria:

* Elective breast surgery due to breast cancer
* Voluntary
* BMI ≥ 18 and ≤ 35 kg/m2
* ASA 1-3
* No regular use of beta-blockers or during the last 72 hours
* No contraindications to beta-blockers

Exclusion Criteria:

* Pregnancy or breast feeding
* AV-block, degree II or III
* Untreated cardiac insufficiency
* Sinus bradycardia, heart rate < 45 / min or symptoms
* Sick sinus syndrome
* Cardiogenic shock
* Severe peripheral vascular disorder
* Systolic blood pressure < 100 mmHg
* Long PQ-time, > 0,24 seconds
* Known hypersensitivity to beta-blockers or the ingredients of the drug

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-03-21 (Estimated); Primary Completion 2018-03-21 (Estimated); Study Completion 2018-03-21 (Estimated)

PRIMARY OUTCOMES:
Anaesthesia | Intraoperative
  Total consumption of desflurane
Anaesthesia | Intraoperative
  Total consumption of remifentanil
Postoperative pain | First 4 postoperative hours
  Total analgesics consumption
Postoperative pain | First 4 postoperative hours
  Time to analgesics
Postoperative pain | First 4 postoperative hours
  Numerical pain scale (0 = no pain, 10 = most pain) at rest and at movement
Long-term pain | 3 months
  The incidence and the level of pain at 3 months
Long-term pain | 1 year
  The incidence and the level of pain at 12 months

SECONDARY OUTCOMES:
Safety and tolerability | Perioperative
  Number of patients with adverse effects
Distribution to the central nervous system | Perioperative
  Cerebro spinal fluid and blood samples
Life satisfaction | 1 year
  Life satisfaction in a Likerts scale
Anxiety | 1 year
  Spielberg State-Trait Anxiety Inventory
Depression | 1 year
  Beck Depression Inventory